CLINICAL TRIAL: NCT02208635
Title: Absorption of Zinc (Zn) From Zn-biofortified and Zn-fortified Maize in Young Zambian Children Between 24-36 Months
Acronym: HPZM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University Teaching Hospital, Lusaka, Zambia (Other); HarvestPlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 14-1126
Record Dates: First submitted 2014-08-01; First posted 2014-08-05 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Nutritional Deficiency
Keywords: Zinc Absorption; Biofortification; Maize; Zambia; Stable isotopes of Zn
MeSH Terms: conditions — Malnutrition; Callosities

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Biofortified Maize (Experimental): Participants in this arm were fed zinc biofortified maize (~30 µg Zn/g).
  Interventions: Other: Biofortified Maize
- Fortified Maize (Experimental): Participants in this arm were fed zinc-oxide fortified maize (total level of ~60 µg Zn/g).
  Interventions: Other: Fortified Maize
- Control Maize (Active Comparator): Participants in this arm were fed maize that was not fortified or biofortified (~15 µg Zn/g maize).
  Interventions: Other: Control Maize

INTERVENTIONS:
Other: Biofortified Maize — Participant in this arm were fed zinc biofortified maize (~30 µg Zn/g).
  Arms: Biofortified Maize
Other: Fortified Maize — Participants in this arm were fed zinc-oxide fortified maize (total level of ~60 µg Zn/g).
  Arms: Fortified Maize
Other: Control Maize — Participants in this arm were fed maize that was not fortified or biofortified (~15 µg Zn/g maize).
  Arms: Control Maize

SUMMARY:
The objective of this study is to compare the quantity of Zn absorbed from an accurately weighed quantity (~100 g) of minimally milled control maize (~15 µg Zn/g maize), from biofortified maize (~30 µg Zn/g) and from the same control maize that has been fortified (total level of ~60 µg Zn/g) when fed to young children age 24-36 months whose major habitual food staple is maize.

DETAILED DESCRIPTION:
Participating children were randomized to receive an accurately weighed quantity of ~100g/day of either the control, fortified or biofortified study maize for 1 day.

On day 1, mothers brought their child to the health center before breakfast. All meals were extrinsically labeled with a zinc stable isotope (70Zn). Meals on this day were consumed in the presence of the research staff. The quantities of nshima or porridge prepared and eaten were accurately weighed and duplicate meals were collected for subsequent mineral analyses.

Between lunch and dinner on day 1 at the Health Center, a blood sample was collected for Hb and plasma Zn analyses and, immediately after and through the same needle, a stable isotope of zinc was intravenously administered into a forearm vein over 1-2 minutes. The family then returned home.

Morning spot urine samples were collected twice daily starting on day 5 and continuing through day 8. Once these collections were finished, the study for this child was complete.

Dietary Zn was measured from laboratory assays of the duplicate test meals. Fractional absorption of Zn (FAZ) was measured by dual isotope tracer ratio methods in urine. Absorbed Zn was calculated by multiplying dietary Zn by FAZ.

ELIGIBILITY:
Inclusion Criteria:

* Children age 24 to 36 months
* Maize meal accounts for at least 75% energy intake
* Able to consume 100 g maize flour/day
* Clinically healthy (stunting is acceptable)
* Lives in target community

Exclusion Criteria:

* Children with chronic or other known chronic disease
* If children are receiving zinc-fortified products, these products will need to be withheld for 2 weeks prior to the study

Ages: 24 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2012-10; Primary Completion 2014-01 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Absorption of zinc | 1 day
  Absorption of zinc will be measured in young children fed a diet of control, Zn-biofortified, or Zn-fortified maize. Fractional absorption of zinc from all meals of the day will be measured by extrinsic labeling with stable isotopes of zinc. Fractional absorption of zinc will be measured by a dual isotope tracer ratio technique. Measurement of total zinc in duplicate diets on test day will allow determination of quantity of this micronutrient absorbed (mg/d).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hambidge, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States
- University Teaching Hospital, Lusaka, Zambia

REFERENCES:
- [Result] Chomba E, Westcott CM, Westcott JE, Mpabalwani EM, Krebs NF, Patinkin ZW, Palacios N, Hambidge KM. Zinc absorption from biofortified maize meets the requirements of young rural Zambian children. J Nutr. 2015 Mar;145(3):514-9. doi: 10.3945/jn.114.204933. Epub 2015 Jan 21. PMID 25733467